CLINICAL TRIAL: NCT05373173
Title: Can a Novel Telemedicine Tool Reduce Disparities Related to the Identification of Preschool
Brief Title: Can a Novel Telemedicine Tool Reduce Disparities Related to the Identification of Preschool Children With Autism?
Acronym: TAP-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Zachary Warren, Professor of Pediatrics; Director of the Division of Developmental Medicine, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 220273; R21MH128790 (NIH)
Record Dates: First submitted 2022-05-05; First posted 2022-05-13 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; ASD; Telehealth; Preschool; Tele-assessment
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-assessment only (Experimental): Families will complete a tele-assessment only.
  Interventions: Behavioral: Tele-assessment only
- Tele-assessment + In-person assessment (Experimental): All families will receive an in-person tele-assessment appointment and an in-person evaluation.
  Interventions: Behavioral: Tele-assessment + In-person assessment

INTERVENTIONS:
Behavioral: Tele-assessment + In-person assessment — All consented families will complete an initial home-based tele-assessment visit via Zoom that includes the TAP-Preschool and a brief symptom-focused developmental interview with a consented clinician. The initial tele-assessment session includes interviewing and developmental assessment to mimic real-world use of TAP-Preschool. After the session, the examiner will record the clinical diagnosis issued (ASD, other developmental concerns, or typical development) and complete two diagnostic certainty ratings. All initial TAP-Preschool administrations will be recorded via Zoom, and 50% of administrations (randomly selected) will be co-scored by a blinded examiner, unaware of prior assessment results and diagnostic decision, to evaluate inter-rater reliability. Within 7 days of the remote assessment, families will participate in an in-person diagnostic assessment including common comprehensive measures of ASD, cognitive skills, and adaptive behavior.
  Arms: Tele-assessment + In-person assessment
Behavioral: Tele-assessment only — Consented families will complete home-based tele-assessment via Zoom that includes the TAP-Preschool. Each participant will have recent data available from comprehensive evaluation tools (ADOS-2, cognitive functioning, adaptive skills). After the session, participating caregivers will provide information about acceptability and challenges.
  Arms: Tele-assessment only

SUMMARY:
Families seeking evaluation for autism spectrum disorder (ASD) often face barriers such as low availability of specialists, lengthy waitlists, and long distances to tertiary care diagnostic centers. This is especially true for children from traditionally underserved groups and communities. Without innovative approaches for enhanced identification of ASD, families and clinicians will continue to struggle with accessing and providing care. Telemedicine offers tremendous potential for addressing this need, but there are few psychometrically sound, validated tools that can be administered remotely, via telehealth platforms. This team of investigators developed and conducted a preliminary evaluation of a novel parent-administered, clinician-guided tele-diagnostic tool, the TAP (TELE-ASD-PEDS), designed specifically for direct-to-home and community clinic use with toddlers. Remote administration of the TAP yielded a very high level of agreement with blinded comprehensive evaluation regarding ASD risk classification. Subsequently, the unanticipated broad dissemination of the TAP during COVID-19 demonstrated its value for traditionally underserved groups, spanning broad geographies. Although promising, this work was limited by its specific focus on toddlers with ASD concerns. A telemedicine tool designed for the unique context and population of preschool-aged children referred for diagnostic assessment could have tremendous value in terms of both accurate identification as well as family engagement with service. In the current work, the investigators will now evaluate the performance, usability, and utility of the TAP-Preschool, a new telemedicine tool for ASD risk assessment in preschoolers, through a clinical trial. The TAP-Preschool was developed through a computationally informed co-production in which the targeted population were recruited as active partners in designing the tool. The investigators will gather critical data not only regarding its structure and accuracy, but also its potential deployment across systems responsible for engaging children and families from underserved groups in meaningful service. This work has potential to transform the ASD evaluation process and dramatically improve care access for traditionally underserved groups.

DETAILED DESCRIPTION:
Innovative telemedicine practices could address many existing traditional barriers to ASD identification. Telemedicine has the potential to put linguistically and culturally competent clinical expert virtual providers directly into communities during a critical window in which many vulnerable families may approach, or re-approach, care systems about developmental concerns that become more prominent with age. In the current proposal, the investigators will evaluate the potential clinical and familial value of a telemedicine-based ASD assessment tool, the TAP-Preschool (TELE-ASD-PEDS-Preschool), designed to overcome traditional barriers to diagnosis and service access in underserved preschool populations that may not be readily identified or engaged by early screening and intervention systems.

A growing body of literature supports the use of telemedicine-based approaches to ASD assessment and intervention. This includes remote activities to assess infant social communication skills in the first year of life, coaching parents through administration of gold standard diagnostic tests, and provider coding and analysis of interactions that are video-recorded by caregivers. Results reflect high levels of caregiver and provider satisfaction and satisfactory agreement with traditional in-person evaluations, illustrating both the promise and feasibility of tele-assessment. However, most existing approaches are limited by a focus on screening rather than diagnosis, protocols requiring specific materials, or asynchronous analysis of submitted videos, which require resources that preclude broader use. Moreover, in current form, these tools are not designed or intended to yield a quantitative formal assessment of core ASD symptoms to support diagnostic decision-making. Further, although providers are increasingly exploring telemedicine approaches to ASD assessment in the context of the COVID-19 pandemic, there is limited published work to date on the use of real-time, caregiver-led ASD assessment in home settings with diverse populations. Prior work from the investigators' team has focused almost exclusively on toddlers in this regard. Ultimately, very few viable tools with validated psychometric properties are available for use in current models of telehealth assessment and care.

In earlier work, we applied machine learning models and the principles of feature engineering to a phenotypically rich clinical research data set of preschoolers with ASD and other developmental concerns (N=914: 594 ASD and 320 Non-ASD) to identify key behavioral targets for tool development. We then engaged in a rigorous adaptation and translation approach to optimize design of the TAP-Preschool. We included leading ASD assessment experts, providers dedicated to caring for underserved populations, and parents of preschool children with ASD from underserved racial/ethnic and linguistic groups. We lead these groups in a collaborative design process in order to yield a set of interactive and play-based, parent-coached tele-assessment activities designed to 1) elicit observations tied to key computational features, 2) be deployed within a 30-minute timeframe, 3) employ inexpensive materials found in most homes, and 4) use accessible assessment instructions for real-time coaching of parents.

The investigators will now deploy the preliminary TAP-Preschool with a small sample (n = 30) to assess acceptability/feasibility, potential clinical value for remote observation, and challenges that warrant revision. These data will then be used to modify the TAP-Preschool and the refined tool will be deployed with a new sample of clinically referred children (n=120). The investigators will evaluate its ability to facilitate accurate telemedicine supported diagnostic decision-making.

Initial deployment, evaluation, and refinement of the TAP-Preschool:

Participants: Investigators will recruit 30 parent/child dyads (children ages 36 to 72 months) with existing diagnoses of ASD (n = 20) or other developmental concerns (n = 10) from a clinical research database. Each participant will have recent data available from comprehensive evaluation tools (ADOS-2, cognitive functioning, adaptive skills). Children with and without ASD are included to provide information about TAP-Preschool usage across diverse phenotypic profiles. The sample size of 30 is deemed adequate for gathering detection of feasibility/acceptability issues and key feedback regarding measure modification for further validation.

Assessment on psychometrics, clinical, and familial value of the TAP-Preschool:

Participants: Investigators will recruit a novel sample (n = 120) parent/child dyads (children 36 - 72 months of age) referred for evaluation of ASD or developmental delays. These children and a primary caregiver will participate in a home-based tele-assessment session and a subsequent blinded in-person evaluation. English/Spanish speaking families with access to a device that will support Zoom will be included.

Initial deployment, evaluation, and refinement of the TAP-Preschool:

Consenting families will be scheduled for a single tele-assessment session with a consented licensed psychologist ("remote clinician") from our clinical research center (n=10). This clinician will coach parents through the TAP-Preschool procedures. Although families will receive standard, basic support regarding tele-assessment procedures, they will not receive extensive training on the TAP-P prior to the session in order to mimic real-world use. All remote clinicians will be experts in ASD with training on the original TAP and ADOS-2 research reliability. Each clinician will participate in 3 sessions (2 children with ASD, 1 other developmental concerns). Clinicians will be blinded to child diagnostic status. Participating telemedicine clinicians in this aim will not be aware of the ratio (2:1 ASD vs. other DD) or recruitment status prior to evaluation ratings. As children will have existing diagnoses, no diagnostic feedback will be provided.

Investigators will collect user data (caregiver, clinicians) on satisfaction, ease of implementation, and diagnostic certainty (clinicians only). Based on this feedback, the preliminary TAP-Preschool instructions and procedures will be modified as needed. To systematically measure acceptability and feasibility of use, investigators will utilize an adapted Acceptability, Likely Effectiveness, Feasibility, and Appropriateness Questionnaire (ALFA-Q).54 The ALFA-Q asks caregivers and clinicians to use a 5-point Likert scale to rate the instrument acceptability, effectiveness, feasibility, and appropriateness for ASD decision making. We will also solicit free-form input. Team leads will briefly interview each clinician and caregiver about their experiences. After each telemedicine evaluation, participating clinicians will view data from previous comprehensive evaluations. Clinicians will provide concrete task evaluation data regarding whether they were able to elicit such behaviors or information in the telemedicine evaluation process. It is important to note that diagnostic agreement rankings will include dichotomous (agree/disagree) and uncertainty data (Likert ratings). As in previous preliminary feasibility/effectiveness trial, investigators will target >60% of providers agreeing with existing risk classification for ASD, <10% of ASD inaccurately identified with ASD, and >50% non ASD DD with certainty as key benchmarks for understanding potential meaningful clinical value. Based on this data, the investigative team will collaborate with the clinical design team to suggest instrument modifications. The tele-assessment will take <45 minutes to complete. The parent forms will take approximately 20 minutes to complete.

Assessment on psychometrics, clinical, and familial value of the TAP-Preschool (Novel Sample):

All consented families will complete an initial home-based tele-assessment visit via Zoom that includes the TAP-Preschool and a brief symptom-focused developmental interview with a consented clinician. The initial tele-assessment session includes interviewing and developmental assessment to mimic real-world use of TAP-Preschool. The visit is designed to take less than 90 minutes, with TAP-Preschool evaluation lasting <30 minutes. All sessions will be timed. After the session, the examiner will record the clinical diagnosis issued (ASD, other developmental concerns, or typical development) and complete two diagnostic certainty ratings, one dichotomous, the other continuous. All initial TAP-Preschool administrations will be recorded via Zoom, and 50% of administrations (randomly selected) will be co-scored by a blinded examiner, unaware of prior assessment results and diagnostic decision, to evaluate inter-rater reliability. Within 7 days of the remote assessment, families will participate in an in-person diagnostic assessment including common comprehensive measures of ASD, cognitive skills, and adaptive behavior. Twenty-five percent of families will be randomly selected to participate in a remote home-based re-test with TAP-Preschool two weeks following initial administration.

Tele-assessment measures: Prior to the appointment, caregivers will complete a Demographics Questionnaire (i.e., age, gender race/ethnicity, zip code, parent education) and a Medical History Form through a secure HIPAA-compliant web portal (REDCap). To reduce technology-related disruptions, research staff will talk to families before the visit about connectivity settings and recommended materials. These will take approximately 20 minutes to complete.

In a single tele-assessment session modeled after our previous work, licensed clinicians will administer the TAP-Preschool, the Developmental Profile, 4th edition (DP-4), and an interview on ASD-related symptoms based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). The DP-4 is a caregiver interview (birth - 21 years) that identifies developmental strengths and weaknesses in five core areas. The DSM-5 interview provides symptom-focused questions with developmental anchors pertinent to this age range. Immediately after the session, the clinician will complete a DSM-5 checklist indicating symptoms present and clinical diagnosis issued (ASD, other developmental concerns, or typical development). This form also contains dichotomous (certain/uncertain) and continuous (10-point Likert scale) certainty ratings. Clinicians will describe their satisfaction with the tele-assessment process (CSQ: Clinician Satisfaction Questionnaire). The initial tele-assessment appointment with the psychologist will last approximately 90 minutes.

Blinded in-person assessment measures: The in-person examiner will be blinded to the tele-assessment diagnosis until after the in-person assessment. The diagnostic confirmation battery will include the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) (one module is chosen based on language ability), a cognitive measure (Mullen Scales of Early Learning or Differential Ability Scales 2nd Edition, the Vineland Adaptive Behavior Scales, Third Edition, and a DSM-5 ASD Interview. Immediately after the in-person session, the examiner will also complete a DSM-5 checklist and certainty ratings. In-person appointments will last approximately 2-3 hours and will consist of traditional diagnostic evaluations for autism spectrum disorder.

Parent measures: Parents will complete the Parent Perceptions of Telehealth (PPT) and the Parent Service Satisfaction (PSS) surveys, used in our previous work, to assess perceptions of tele-assessment procedures after the telemedicine and in-person evaluations. These parent forms will take approximately 10 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Initial deployment (n = 30):
* English/Spanish Speaking families
* Children 36-72 months of age
* access to a device capable of supporting Zoom
* already has participated in a diagnostic evaluation

Novel sample (n = 120):

Inclusion

* English/Spanish Speaking families
* Children 36-72 months of age
* access to a device capable of supporting Zoom
* has not participated in a diagnostic evaluation

Exclusion Criteria:

* Initial deployment (n = 30):
* severe sensorimotor impairments

Novel sample (n = 120):

- severe sensorimotor impairments

Ages: 36 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Warren, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner L, Vehorn A, Weitlauf AS, Lavanderos AM, Wade J, Corona L, Warren Z. Development of a Novel Telemedicine Tool to Reduce Disparities Related to the Identification of Preschool Children with Autism. J Autism Dev Disord. 2025 Jan;55(1):30-42. doi: 10.1007/s10803-023-06176-3. Epub 2023 Dec 8. PMID 38064003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Children were recruited together with a participating primary caregiver (i.e., parent-child dyads). Study sample size below and throughout results is reflective of parent-child dyads.
Groups:
- Tele-assessment Only: Each parent-child dyad will complete a tele-assessment only. Consented dyads will complete home-based tele-assessment via Zoom that includes the TAP-Preschool. Each participant will have recent data available from comprehensive evaluation tools (ADOS-2, cognitive functioning, adaptive skills).
- Tele-assessment + In-person Assessment: Each parent-child dyad will receive an in-person tele-assessment appointment and an in-person evaluation. All dyads will participate in an initial home-based tele-assessment visit via Zoom that includes the TAP-Preschool and a brief symptom-focused developmental interview with a consented clinician. The initial tele-assessment session includes interviewing and developmental assessment to mimic real-world use of TAP-Preschool. After the session, the examiner will record the clinical diagnosis issued (ASD, other developmental concerns, or typical development) and complete two diagnostic certainty ratings. All initial TAP-Preschool administrations will be recorded via Zoom, and 50% of administrations (randomly selected) will be co-scored by a blinded examiner, unaware of prior assessment results and diagnostic decision, to evaluate inter-rater reliability. Within 7 days of the remote assessment, dyads will participate in an in-person diagnostic assessment including common comprehensive measures of ASD, cognitive skills, and adaptive behavior.
Period: Overall Study
Arm/Group | Tele-assessment Only | Tele-assessment + In-person Assessment
Started | 30 (Reflects 30 parent-child dyads) | 118 (Reflects 118 parent-child dyads)
Completed | 30 (Reflects 30 parent-child dyads) | 116 (116 parent-child dyads)
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline data are reported separately for child and parent members of each parent-child dyad. Baseline characteristics were not collected for parent participants in the tele-assessment only arm. Age was not collected for parent in either arm.
Groups:
- Tele-assessment Only - Children; Tele-assessment Only - Parents: Each parent-child dyad will complete a tele-assessment only. Consented dyads will complete home-based tele-assessment via Zoom that includes the TAP-Preschool. Each participant will have recent data available from comprehensive evaluation tools (ADOS-2, cognitive functioning, adaptive skills). After the session, participating caregivers will provide information about acceptability and challenges.
- Tele-assessment + In-person Assessment - Children; Tele-assessment + In-person Assessment - Parents: Each parent-child dyad will receive an in-person tele-assessment appointment and an in-person evaluation. All consented dyads will complete an initial home-based tele-assessment visit via Zoom that includes the TAP-Preschool and a brief symptom-focused developmental interview with a consented clinician. The initial tele-assessment session includes interviewing and developmental assessment to mimic real-world use of TAP-Preschool. After the session, the examiner will record the clinical diagnosis issued (ASD, other developmental concerns, or typical development) and complete two diagnostic certainty ratings. All initial TAP-Preschool administrations will be recorded via Zoom, and 50% of administrations (randomly selected) will be co-scored by a blinded examiner, unaware of prior assessment results and diagnostic decision, to evaluate inter-rater reliability. Within 7 days of the remote assessment, dyads will participate in an in-person diagnostic assessment including common comprehensive measures of ASD, cognitive skills, and adaptive behavior.
- Total: Total of all reporting groups
Arm/Group | Tele-assessment Only - Children | Tele-assessment + In-person Assessment - Children | Tele-assessment Only - Parents | Tele-assessment + In-person Assessment - Parents | Total
Number analyzed (Participants) | 30 | 118 | 30 | 118 | 296
Age, Continuous [Mean (Standard Deviation); unit: months] — Population: Age was not collected for parent participants
  months
    number analyzed (Participants) | 30 | 118 | 0 | 0 | 148
    (all) | 49.3 (9) | 47.8 (9.9) |  |  | 47.82 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics were not collected for parent participants in the Tele-assessment only arm. 4 parents in the tele-assessment + in-person arm opted not to report their gender.
  Participants
    number analyzed (Participants) | 30 | 118 | 0 | 114 | 262
    Female | 7 | 33 |  | 102 | 142
    Male | 23 | 85 |  | 12 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics were not collected for parent participants in the tele-assessment only arm. 6 parents in the tele-assessment + in-person arm opted not to provide information about their ethnicity.
  Participants
    number analyzed (Participants) | 30 | 118 | 0 | 118 | 266
    Hispanic or Latino | 9 | 10 |  | 7 | 26
    Not Hispanic or Latino | 21 | 105 |  | 105 | 231
    Unknown or Not Reported | 0 | 3 |  | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics were not collected for parent participants in the tele-assessment only arm. 8 parents in the tele-assessment + in-person arm opted not to provide information about their race.
  Participants
    number analyzed (Participants) | 30 | 118 | 0 | 118 | 266
    American Indian or Alaska Native | 0 | 0 |  | 0 | 0
    Asian | 1 | 4 |  | 6 | 11
    Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0 | 0
    Black or African American | 5 | 23 |  | 21 | 49
    White | 23 | 70 |  | 80 | 173
    More than one race | 1 | 15 |  | 3 | 19
    Unknown or Not Reported | 0 | 6 |  | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 30 | 118 | 30 | 118 | 296

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Certainty: Tele-assessment
Description: Clinicians rated diagnostic certainty on a 4-point Likert Scale. Possible scores range from 1 to 4, with 1 indicating "Completely Uncertain," 2 indicating "Somewhat Uncertain," 3 indicating "Somewhat Certain" and 4 indicating "Completely Certain." Higher values reflect stronger clinician diagnostic certainty.
Time Frame: Single timepoint: Immediately after completing tele-assessment, an average of 90 minutes
Population: Diagnostic certainty is analyzed for child participants only.
Measure: Mean (Standard Deviation); unit: score on a scale (range 1-4)
Groups:
- Tele-assessment Only: Each parent-child dyad will complete a tele-assessment only. Consented dyads will complete home-based tele-assessment via Zoom that includes the TAP-Preschool. Each participant will have recent data available from comprehensive evaluation tools (ADOS-2, cognitive functioning, adaptive skills). After the session, participating caregivers will provide information about acceptability and challenges.
- Tele-assessment + In-person Assessment: Each parent-child dyad will receive an in-person tele-assessment appointment and an in-person evaluation. All consented dyads will complete an initial home-based tele-assessment visit via Zoom that includes the TAP-Preschool and a brief symptom-focused developmental interview with a consented clinician. The initial tele-assessment session includes interviewing and developmental assessment to mimic real-world use of TAP-Preschool. After the session, the examiner will record the clinical diagnosis issued (ASD, other developmental concerns, or typical development) and complete two diagnostic certainty ratings. All initial TAP-Preschool administrations will be recorded via Zoom, and 50% of administrations (randomly selected) will be co-scored by a blinded examiner, unaware of prior assessment results and diagnostic decision, to evaluate inter-rater reliability. Within 7 days of the remote assessment, dyads will participate in an in-person diagnostic assessment including common comprehensive measures of ASD, cognitive skills, and adaptive behavior.
Arm/Group | Tele-assessment Only | Tele-assessment + In-person Assessment
Number analyzed (Participants) | 30 | 116
score on a scale (range 1-4) | 3.07 (0.83) | 2.85 (0.99)

2. Primary Outcome: Family Satisfaction
Description: Parents will complete the Parent Perceptions of Telehealth survey to assess perceptions of tele-assessment procedures. The survey includes seven questions with three response options per questions (Very True, Somewhat True, Not True). The percentage of parents endorsing "very true" is reported.
Time Frame: Single timepoint: Immediately after completing tele-assessment, an average of 90 minutes
Population: In the tele-assessment only group, 27/30 participating parents completed the post-telehealth visit satisfaction survey. In the tele-assessment + in-person assessment group, 114/118 participating parents completed the post-telehealth visit satisfaction survey. Only parents completed satisfaction surveys.
Measure: Number; unit: percentage endorsing "very true"
Groups:
- Tele-assessment Only: Families will complete a tele-assessment only. Consented families will complete home-based tele-assessment via Zoom that includes the TAP-Preschool. Each participant will have recent data available from comprehensive evaluation tools (ADOS-2, cognitive functioning, adaptive skills). After the session, participating caregivers will provide information about acceptability and challenges.
- Tele-assessment + In-person Assessment: All families will receive an in-person tele-assessment appointment and an in-person evaluation. All consented families will complete an initial home-based tele-assessment visit via Zoom that includes the TAP-Preschool and a brief symptom-focused developmental interview with a consented clinician. The initial tele-assessment session includes interviewing and developmental assessment to mimic real-world use of TAP-Preschool. After the session, the examiner will record the clinical diagnosis issued (ASD, other developmental concerns, or typical development) and complete two diagnostic certainty ratings. All initial TAP-Preschool administrations will be recorded via Zoom, and 50% of administrations (randomly selected) will be co-scored by a blinded examiner, unaware of prior assessment results and diagnostic decision, to evaluate inter-rater reliability. Within 7 days of the remote assessment, families will participate in an in-person diagnostic assessment including common comprehensive measures of ASD, cognitive skills, and adaptive behavior.
Arm/Group | Tele-assessment Only | Tele-assessment + In-person Assessment
Number analyzed (Participants) | 27 | 114
percentage endorsing "very true"
  Before I started my child's telehealth visit, I understood what I would be doing. | 96.3 | 93.0
  The instructions the psychologist gave me abouthow to play with my child were easy to follow. | 96.3 | 98.2
  The activities got my child to show the behaviors I am concerned about. | 38.5 | 51.8
  I felt comfortable receiving feedback about my child over telehealth. | 92.6 | 95.6
  The telehealth visit lasted the right amount of time. | 77.8 | 91.2
  I would recommend participating in this kind of telehealth evaluation to others. | 81.5 | 90.4
  The telehealth technology was easy to use. | 100 | 91.9

3. Primary Outcome: Diagnostic Certainty: In-person Assessment
Description: as for outcome 1
Time Frame: Single timepoint: Immediately after completing tele-assessment, an average of 180 minutes
Population: Participants in the Tele-assessment only arm did not receive in-person assessment. Diagnostic certainty is analyzed for child participants only.
Measure: Mean (Standard Deviation); unit: score on a scale (range 1-4)
Arm/Group | Tele-assessment Only | Tele-assessment + In-person Assessment
Number analyzed (Participants) | 0 | 116
score on a scale (range 1-4) |  | 3.64 (0.67)

4. Primary Outcome: Diagnostic Accuracy of TAP-P
Description: For the preliminary tele-assessment only arm, diagnostic accuracy reflects the percentage of participants for whom the tele-assessment clinician's diagnostic impression (autism vs not autism) was in agreement with the child's existing diagnosis (autism vs not autism).
  For the tele-assessment + in-person assessment arm, diagnostic accuracy reflects the percentage of participants for whom the tele-assessment clinician's diagnostic impression (autism vs not autism) was in agreement with the diagnostic determination following in-person assessment (autism vs not autism).
Time Frame: Single timepoint: Calculated immediately after completion of in-person assessment
Population: Diagnostic accuracy is calculated for child participants only.
Measure: Number; unit: percentage of participants
Arm/Group | Tele-assessment Only | Tele-assessment + In-person Assessment
Number analyzed (Participants) | 30 | 116
percentage of participants | 60 | 81.9

ADVERSE EVENTS:
Time Frame: Day of assessment
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Tele-assessment Only - Children; Tele-assessment Only - Parents: Parent-child dyads will complete a tele-assessment only.
  Tele-assessment only: Consented dyads will complete home-based tele-assessment via Zoom that includes the TAP-Preschool. Each participating child will have recent data available from comprehensive evaluation tools (ADOS-2, cognitive functioning, adaptive skills). After the session, participating caregivers will provide information about acceptability and challenges.
- Tele-assessment + In-person Assessment - Children; Tele-assessment + In-person Assessment - Parents: Parent-child dyads will complete a tele-assessment appointment and an in-person evaluation.
  Tele-assessment + In-person assessment: All consented dyads will complete an initial home-based tele-assessment visit via Zoom that includes the TAP-Preschool and a brief symptom-focused developmental interview with a consented clinician. The initial tele-assessment session includes interviewing and developmental assessment to mimic real-world use of TAP-Preschool. After the session, the examiner will record the clinical diagnosis issued (ASD, other developmental concerns, or typical development) and complete two diagnostic certainty ratings. All initial TAP-Preschool administrations will be recorded via Zoom, and 50% of administrations (randomly selected) will be co-scored by a blinded examiner, unaware of prior assessment results and diagnostic decision, to evaluate inter-rater reliability. Within 7 days of the remote assessment, dyads will participate in an in-person diagnostic assessment including common comprehensive measures of ASD, cognitive skills, and adaptive behavior.
Arm/Group | Tele-assessment Only - Children | Tele-assessment + In-person Assessment - Children | Tele-assessment Only - Parents | Tele-assessment + In-person Assessment - Parents
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/118 | 0/30 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/118 | 0/30 | 0/118
Other Adverse Events (participants affected / at risk) | 0/30 | 0/118 | 0/30 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT05373173/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT05373173/ICF_000.pdf